CLINICAL TRIAL: NCT00344175
Title: Double-blind follow-on Study of Pitavastatin (4mg) Versus Simvastatin (40mg and 80mg) With a Single-blind Extension of Treatment in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia and 2 or More Risk Factors for Coronary Heart Disease
Brief Title: Follow-on Protocol of Pitavastatin Versus Simvastatin in Patients With Hypercholesterolemia or Dyslipidemia and Coronary Heart Disease Risk Factors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Dragos Budinski, Kowa Research Europe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK-104-309
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia; Dyslipidemia; Coronary Heart Disease
Keywords: hypercholesterolemia; dyslipidemia; CHD; pitavastatin; simvastatin; 2 or more risk factors for coronary heart disease; combined dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Coronary Disease | interventions — pitavastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 4 mg (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: pitavastatin
- Simvastatin 40mg/80mg (Active Comparator): Simvastatin 40 mg or 80 mg once daily
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: pitavastatin
  Arms: Pitavastatin 4 mg
Drug: simvastatin
  Arms: Simvastatin 40mg/80mg

SUMMARY:
This is a sixteen-week follow-on and 28 week single-blind extension study for patients who participated in study NK-104-304.

DETAILED DESCRIPTION:
This is a sixteen-week, double-blind, active controlled, follow-on and 28 week single blind extension study for patients who participated in NK-104-304.

ELIGIBILITY:
Inclusion Criteria:

* Completed NK-104-304 (NCT 00309738)
* Hypercholesterolemia or combined dyslipidemia
* 2 or more risk factors for coronary heart disease (CHD)

Exclusion Criteria:

* Withdrawn or terminated from NK-104-304 (00309738)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, MD, Study Director — Kowa Research Europe
Locations (28):
- Denmark (4):
  - Y Forskning, Bispebjerg Hospital, Copenhagen Nv
  - Frederiks Hospital, Kardiologisk, Frederiksberg
  - Kolesterollaboratoriet, Hellerup
  - CCBR A/S, Vejle
- Netherlands (8):
  - Middellaan 5, Breda
  - Bomanshof 8, Eindhoven
  - Damsterdiep 9, Groningen
  - Doezastraat 1, Leiden
  - Kamerlingh Onnesstraat 16-18, Nijmegen
  - Mathenesserlaan 247, Rotterdam
  - Reigerstraat 30, Velp
  - Parkdreef 142, Zoetermeer
- Spain (6):
  - Hospital Clinico S. Juan de Alicante, San Juan, Alicante
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- Sweden (10):
  - Angelholms Sjukhus, Medicinkliniken, Angelhom
  - Sahlgrenska University Hospital, Intermedicin, Gothenburg
  - Hjartmottagningen, Helsingborg
  - Lakarcentrum Nyponet, Karineholm
  - Medicinkliniken, Ludvika
  - Huslakaren i Sandviken, Sandviken
  - Narsjukhuset Sandviken, Kardiologlab, Medicin, Sandviken
  - Hjart & Karlcenter, Södertälje
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjarthuset AB, Varberg

REFERENCES:
- [Derived] Eriksson M, Budinski D, Hounslow N. Long-term efficacy of pitavastatin versus simvastatin. Adv Ther. 2011 Sep;28(9):799-810. doi: 10.1007/s12325-011-0057-6. Epub 2011 Aug 25. PMID 21874537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with primary hypercholesterolemia or combined dyslipidemia, who have satisfied the inclusion/exclusion criteria of the core study, and completed the core study were eligible for this study.
Groups:
- Pitavastatin 4 mg: Ptavastatin 4 mg once daily
Period: Overall Study
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg
Started | 121 | 57
Completed | 109 | 47
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg | Total
Number analyzed (Participants) | 121 | 57 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 44 | 142
  >=65 years | 23 | 13 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (5.80) | 60.8 (6.52) | 60.5 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 18 | 57
  Male | 82 | 39 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Attaining NCEP LDL-C Target at Week 16
Description: Number of patients attaining the National Cholesterol Education Program (NCEP) LDL-C target at Week 16. According to NCEP criteria the target LDL-C is 100 mg/dL.
Time Frame: 16 weeks
Population: All patients who received at least 1 dose of study drug and who had at least 1 on-treatment (post Visit 1) lipid assessment.
Measure: Number; unit: particpants
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg
Number analyzed (Participants) | 108 | 52
particpants | 98 | 45

2. Primary Outcome: Number of Patients Attaining NCEP LDL-C Target at Week 44
Description: Number of patients attaining National Cholesterol Education Program (NCEP) LDL-C target at Week 44. According to NCEP criteria the target LDL-C is 100 mg/dL.
Time Frame: 44 Weeks
Measure: Number; unit: Participants
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg
Number analyzed (Participants) | 108 | 52
Participants | 94 | 42

3. Secondary Outcome: Percent Change From Baseline in LDL-C
Time Frame: Baseline to 44 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg
Number analyzed (Participants) | 108 | 52
percent change | -41.81 (15.130) | -41.37 (16.425)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg | Simvastatin 40mg/80mg
Serious Adverse Events (participants affected / at risk) | 4/121 | 7/57
Other Adverse Events (participants affected / at risk) | 57/121 | 38/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg (N=121) | Simvastatin 40mg/80mg (N=57)
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Global amnesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg (N=121) | Simvastatin 40mg/80mg (N=57)
Nasopharyngitis (Infections and infestations) | 24 | 15
Influenza (Infections and infestations) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1
Headache (Nervous system disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days